CLINICAL TRIAL: NCT06083090
Title: Effects of Yoga Therapy in Rehabilitation Compared to Physiotherapy in Moderate Axial Spondyloarthritis (axSPA): a Randomized Controlled Multicenter Study.
Brief Title: Effects of Yoga Therapy in Rehabilitation Compared to Physiotherapy in Moderate Axial Spondyloarthritis (axSPA)
Acronym: YOKISPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP210998
Record Dates: First submitted 2023-07-21; First posted 2023-10-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Axial Spondyloarthritis (axSPA)
Keywords: Yogatherapy; Ankylosing Spondyloarthritis; Physiotherapy; Yoga; Rheumatism
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Rheumatic Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Multicenter, comparative, randomized study in two parallel groups (yogatherapy versus physiotherapy), of superiority.
Who Masked: Outcomes Assessor
Masking Description: The evaluators of the secondary endpoints relating to measurements of respiratory and biomechanical parameters will be blinded to the patient randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yogatherapy (Experimental): Randomization of 36 patients in the yogatherapy group.
  Interventions: Procedure: Yogatherapy
- Physiotherapy (Active Comparator): Randomization of 36 patients in the physiotherapy group.
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Yogatherapy — The experimental arm will benefit from support by a physiotherapist trained in yoga, in a group for ten weeks with two weekly sessions of approximately 1 hour each. A new yoga program adapted for the axSPA will be implemented.
  Arms: Yogatherapy
Procedure: Physiotherapy — The comparator arm will benefit from support by a physiotherapist, in groups for ten weeks at the rate of two weekly sessions of approximately 1 hour each. An already existing program adapted for the axSPA will be implemented.
  Arms: Physiotherapy

SUMMARY:
A few studies have evaluated the effectiveness of yoga therapy in patients with axial spondyloarthritis (axSPA). On the other hand, studies conducted in other chronic rheumatisms such as low back pain, rheumatoid arthritis or other conditions such as cancer have shown that yogatherapy can have a effective action on the physical and psychological level.

Yogatherapy is a non-drug "body-mind" approach that would be likely to improve the physical symptoms (pain, stiffness, in particular spinal and pelvic), internal organs (colitis) and psychological symptoms as well as the perception of fatigue of people with axSPA. A 2021 study showed the feasibility and acceptability of regular yogatherapy practice in patients with axSPA.

It is therefore necessary to conduct randomized controlled studies to assess the effectiveness of this management strategy.

DETAILED DESCRIPTION:
The term axial spondyloarthritis (axSPA) encompasses various inflammatory diseases of the spine, including ankylosing spondyloarthritis (AS) and non-radiographic axial spondyloarthritis (nr-axSPA).

axSPA is a chronic inflammatory joint disease affecting the axial skeleton. It is the second cause of chronic inflammatory rheumatism and affects 0.5 to 2% of the general population. It generally affects young adults, with a male predominance (2 men for 1 woman).

axSPA can lead to physical consequences (fatigue, pain, stiffness, with in particular serious damage to the spine causing functional impairment, etc.) and psychological consequences (anxiety, depression). It is responsible for a disability and a mediocre quality of life with, moreover, a significant socio-economic impact. In France, it is one of the long-term illnesses and may require heavy treatment.

The medicinal therapeutic side, taken care of by rheumatologists specializing in this pathology, has evolved a lot (from non-steroidal anti-inflammatory drugs [NSAIDs] to anti-tumor necrosis factor [anti-TNF] and anti-interleukin 17 [anti-IL 17]), allowing notable improvements. It is now a question of also developing the non-drug therapeutic side, to contribute to improving the quality of life, thus meeting the demand of patients with chronic diseases.

Information and therapeutic education occupy an important place, with results in favor of an improvement in the management of these diseases.

The recommendations emphasize that the non-pharmacological treatment of axSPA should include regular physical exercise, that individual and group physical therapy sessions should be considered as well as self-exercises.

Several randomized controlled trials have shown that physical therapy with various modalities has positive effects on pain and AS function. Physical therapy therefore also seems to play an important role in the management of patients. It prevents stiffness and improves functional capacity and quality of life.

Physical therapy should be initiated as soon as axSPA is diagnosed and regular exercise should form the basis of management. The review by Zochling et al. as well as a systematic review showed that exercises have positive effects on BASFI, BASDAI functions, pain and mobility. A Cochrane review on the role of physiotherapy interventions in SPA also concluded that physical therapy was beneficial. Physical activity, self-exercises and physiotherapy are part of the 2022 recommendations of the French Society of Rheumatology. Beneficial effects on disease activity were observed in axSPA, with good tolerance for intense exercise.

Recently an Indian team evaluated the effectiveness of online yogatherapy with 60 min structured modules on patients with axSPA for 3 months, with a significant improvement in the BASDAI score.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking patient aged 18 and over
* Patient with axial spondyloarthritis (axSPA) according to Assessment of SpondyloArthritis International Society, diagnosed by a rheumatologist
* "Moderately active" to "active" form of axSPA (basic BASDAI > 3)
* Stable disease: No recent or foreseeable introduction in the next 6 months of drug treatments for axSPA (excluding analgesics)
* Absence of disabling stress urinary incontinence
* Geographical or organizational possibility of undergoing the study
* Patient informed and having signed the informed consent form for participation in the research

Exclusion Criteria:

* Pregnancy or breastfeeding
* Recent childbirth (within the last six months)
* Patient already practicing yoga or having practiced it in the last six months
* Abdominal or spinal surgery in the last six months
* Motor neurological deficit
* Sphincter deficit
* Any other somatic pathology preventing the practice of physiotherapy or yogatherapy according to the opinion of the evaluating clinician
* Depressive syndrome requiring specific treatment
* Non-affiliation to a social security scheme (beneficiary or beneficiary) or to another social protection scheme
* Patient deprived of liberty by judicial or administrative decision or under legal protection (guardianship, safeguard of justice)
* Currently participating in or in a period of exclusion from: another interventional research involving human participants, a clinical trial on a medical product for human, a clinical investigation on a medical device. Participation in non-interventional research is authorized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2028-02-06 (Estimated); Study Completion 2028-08-27 (Estimated)

PRIMARY OUTCOMES:
Evolution of the axSPA global activity score (fatigue, pain, stiffness) | Between the 2 month visit and the 5 month visit.
  Change in the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) score, via a self-administered questionnaire that assesses the "activity" of the disease (6 items, max score = 100, the higher the score the more disabling the disease).

SECONDARY OUTCOMES:
Evolution of the axSPA global activity score (fatigue, pain, stiffness) | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) score, via a self-administered questionnaire that assesses the "activity" of the disease (6 items, max score = 100, the higher the score the more disabling the disease).
Functional impact | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in self-assessment of functional capacity during daily tasks via the BASFI score (Bath Ankylosing Spondylitis disease Functional Index) (10 items, max score = 10, the higher the score the more disabling the disease).
Health-related quality of life | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in the patient's self-assessment via the generic SF-36 scale (Short Form-36 scale) (36 items, max score = 100, the higher the score the better the perception of quality of life).
Anxiety and depression | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in the patient's self-assessment via the HAD scale (Hospital Anxiety and Depression scale) (14 items, max anxiety score = 21, max depression score = 21, the higher the score the more anxiety and depressive disorders are marked).
Respiratory capacity | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Measurement of chest expansion.
Spinal and axial mobility (maximum active amplitudes - sagittal plane) | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in measurement of maximum active amplitudes in orthostatism of the thoraco-lumbar spine in the sagittal (flexion/extension) plane.
Spinal and axial mobility (degrees of kyphosis and lordosis) | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in measurement of the degrees of kyphosis and lordosis while standing.
Spinal and axial mobility (maximum active amplitudes - frontal plane) | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in measurement of maximum active amplitudes in orthostatism of the thoraco-lumbar spine in the frontal (lateral inclinations) plane.
Spinal and axial mobility (podobarometric treadmill) | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in measurement of the spatiotemporal analysis of gait on a podobarometric treadmill.
Axial mobility | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in BASMI (Bath Ankylosing Spondylitis Metrology Index) score (5 items, max score = 10, the higher the score the more restricted the axial mobility).
Follow-up of the therapeutic strategy | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in therapeutic strategy.
Drug consumption monitoring | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in drug consumption.
Sleep quality | Between the 2 month visit and the 5 month visit. Between the 2 month visit and the 11 month visit.
  Change in QESL score (Leeds Sleep Assessment Questionnaire) (10 visual analog scales, minimum = -50, maximum = 50, the higher the score the better the sleep).
Adherence to the practice of yogatherapy of patients randomized in this group | After physical rehabilitation : at 5 month and 11 month visits.
  Degree of adherence to the practice of yogatherapy collected through responses to a short self-questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Petra PAREJO MARGALLO, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital Avicenne, Bobigny
  - Hôpital Henri Mondor, Créteil
  - Hôpital Pitié Salpetrière, Paris
  - Hôpital Cochin, Paris

IPD SHARING:
Plan to Share IPD: No
Datas are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information.